CLINICAL TRIAL: NCT01862614
Title: A Prospective Randomized, Double-blind Study of the Anesthetic Efficacy of Buffered Articaine as a Primary Buccal Infiltration of the Mandibular First Molar.
Brief Title: Testing the Anesthetic Effectiveness of Buffered Articaine Injected Next to a Lower First Molar.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, John Nusstein, Professor, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Buffered Articaine
Record Dates: First submitted 2013-05-22; First posted 2013-05-24 (Estimated); Results first posted 2020-12-02 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Anesthetic Effectiveness
Keywords: Degree of pulpal anesthesia obtained.; Primary infiltration in the lower first molar.; Buffered local anesthetic.
MeSH Terms: interventions — Carticaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Buffered Articaine at 1st Appointment (Experimental): Subjects received an infiltration injection of 1.8cc buffered 4% articaine.
  Interventions: Drug: Buffered Articaine Hydrochloride + Epinephrine
- Articaine at 1st Appointment (Active Comparator): Subjects received an infiltration injection of 1.8cc 4% articaine (unbuffered).
  Interventions: Drug: Articaine Hydrochloride + Epinephrine

INTERVENTIONS:
Drug: Articaine Hydrochloride + Epinephrine
  Arms: Articaine at 1st Appointment
Drug: Buffered Articaine Hydrochloride + Epinephrine
  Arms: Buffered Articaine at 1st Appointment

SUMMARY:
Infiltration (injecting next to the tooth) injections are common in dentistry and a number of studies have shown that articaine anesthetic, when injected next to a lower molar, is more effective than a local anesthetic injection of lidocaine. However success rates have not been as high as hoped for. No objective study has addressed the success rate of buffering articaine in a mandibular primary buccal infiltration of the first molar. Therefore, the purpose of this prospective, randomized, double-blind, crossover study is to compare the degree of pulpal anesthesia obtained with a buffered 4% articaine with 1:100,000 epinephrine solution versus a non-buffered 4% articaine with 1:100,000 epinephrine solution as a primary infiltration in the mandibular first molar. The investigators will also record the pain of injection and postoperative pain.

DETAILED DESCRIPTION:
Using a crossover design, 80 adult subjects will receive two injections consisting of a primary mandibular first molar infiltration of 1.8 mL of non-buffered 4% articaine with 1:100,000 epinephrine, and 1.8 mL of buffered 4% articaine with 1:100,000 in two separate appointments spaced at least one week apart. With the crossover design, 160 infiltrations will be given for the first molar and each subject will serve as his or her own control. Eighty infiltrations will be administered on the mandibular left side and 80 administered on the mandibular right side. The order of the two injections will be assigned randomly and the dentist and subject will be blinded about which anesthetic the subject is given. The anesthetics used in this study are not experimental. An electric pulp tester (EPT) will be used to test the lower first molar for anesthesia starting 30 seconds after the injection; and testing every 30 seconds for the first five minutes. After five minutes the EPT will be used to test the lower first molar every minute and the contralateral control canine every 5 minutes for a grand total of sixty minutes. The pain of injection and postoperative pain will be recorded in a survey. Patients will report any postoperative pain or discomfort on a Visual Analog Scale (VAS) for three days following each appointment. The data will be statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Between the age of 18-65 years.
* in good health (ASA classification II or higher).
* able to provide informed consent.

Exclusion Criteria:

* allergy to articaine.
* history of significant medical problems (ASA classification of III or worse).
* diagnosed depression (taking tri-cyclic antidepressant medications to control).
* have taken central nervous system (CNS) depressants (including alcohol or any analgesic medications) within the last 48 hours prior to testing.
* lactating or pregnant.
* inability to give informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University College of Dentistry, Postle Hall, Columbus, Ohio, United States

REFERENCES:
- [Background] Kanaa MD, Whitworth JM, Corbett IP, Meechan JG. Articaine and lidocaine mandibular buccal infiltration anesthesia: a prospective randomized double-blind cross-over study. J Endod. 2006 Apr;32(4):296-8. doi: 10.1016/j.joen.2005.09.016. Epub 2006 Feb 17. PMID 16554198
- [Background] Robertson D, Nusstein J, Reader A, Beck M, McCartney M. The anesthetic efficacy of articaine in buccal infiltration of mandibular posterior teeth. J Am Dent Assoc. 2007 Aug;138(8):1104-12. doi: 10.14219/jada.archive.2007.0324. PMID 17670879
- [Background] Corbett IP, Kanaa MD, Whitworth JM, Meechan JG. Articaine infiltration for anesthesia of mandibular first molars. J Endod. 2008 May;34(5):514-8. doi: 10.1016/j.joen.2008.02.042. PMID 18436027
- [Background] Abdulwahab M, Boynes S, Moore P, Seifikar S, Al-Jazzaf A, Alshuraidah A, Zovko J, Close J. The efficacy of six local anesthetic formulations used for posterior mandibular buccal infiltration anesthesia. J Am Dent Assoc. 2009 Aug;140(8):1018-24. doi: 10.14219/jada.archive.2009.0313. PMID 19654255
- [Background] Sinnott CJ, Garfield JM, Thalhammer JG, Strichartz GR. Addition of sodium bicarbonate to lidocaine decreases the duration of peripheral nerve block in the rat. Anesthesiology. 2000 Oct;93(4):1045-52. doi: 10.1097/00000542-200010000-00028. PMID 11020760
- [Background] Burmeister CH. A practical method for the extemporaneous preparations of a buffered anesthetic solution. J Am Dent Assoc 22:1514, 1935.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 80 subjects will be recruited in this crossover study. Each of the subjects will receive the injection regimens at 2 separate appointments spaced at least 2 weeks apart.
Groups:
- Articaine (First): Subjects receiving 1.8cc articaine injection at first appointment.
- Buffered Articaine (First): Subjects receiving injection of 1.8cc buffered articaine at first appointment.
Period: First Appointment.
Arm/Group | Articaine (First) | Buffered Articaine (First)
Started | 40 (Received articaine injection at first appointment.) | 40 (Received buffered articaine at first appointment.)
Completed | 40 | 40
Not Completed | 0 | 0
Period: 2 Week Washout Period.
Arm/Group | Articaine (First) | Buffered Articaine (First)
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0
Period: Second Appointment.
Arm/Group | Articaine (First) | Buffered Articaine (First)
Started (Received buffered articaine at second appointment.) | 40 (Received buffered articaine at second appointment.) | 40 (Received articaine at second appointment.)
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Articaine: Subjects receiving articaine injection.
Arm/Group | Articaine
Number analyzed (Participants) | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 80
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.3 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 42
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 80

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving Pulpal Anesthesia.
Description: An electric pulp tester will be used to test the lower jaw teeth (molars, premolars, and incisors) for anesthesia (numbness) in 4-minute time cycles for 60 minutes. Measurements of less than 80 on the EPT is considered not numb (anesthesia failure). Readings of 80 equate to anesthetic success.
Time Frame: 60 minutes per injection sequence.
Measure: Count of Participants; unit: Participants
Groups:
- Buffered Articaine: Subjects receiving an injection of 1.8cc buffered articaine.
Arm/Group | Articaine | Buffered Articaine
Number analyzed (Participants) | 80 | 80
Participants | 52 | 57

ADVERSE EVENTS:
Groups:
- Articaine: Subjects receiving injection of 1.8cc 4% articaine.
- Buffered Articaine: Subjects receiving injection of 1.8cc buffered 4% articaine.
Arm/Group | Articaine | Buffered Articaine
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/80
Other Adverse Events (participants affected / at risk) | 0/80 | 0/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No